CLINICAL TRIAL: NCT06438887
Title: Strategic Ingestion of Creatine Supplementation and Resistance Training in Trained Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Principal Investigator, Darren Candow, Professor, University of Regina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio-REB 4641
Record Dates: First submitted 2024-05-16; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Strength; Muscle
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Creatine Before Training (Experimental): 5 grams of creatine monohydrate + 3 grams of placebo immediately before training sessions; 8 grams of placebo immediately after training sessions; 8 grams of placebo on non-training days.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Creatine monohydrate
- Creatine After Training (Experimental): 5 grams of creatine monohydrate + 3 grams of placebo immediately after training sessions; 8 grams of placebo immediately before training sessions; 8 grams of placebo on non-training days.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Creatine monohydrate
- Creatine Non-Training (Experimental): 5 grams of creatine monohydrate + 3 grams of placebo on non-training days; 8 grams of placebo immediately before training sessions; 8 grams of placebo immediately after training sessions.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): 8 grams of placebo immediately before training sessions; 8 grams of placebo immediately after training sessions; 8 grams of placebo on non-training days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Corn-Starch Maltodextrin
Dietary Supplement: Creatine monohydrate — Creatine
  Arms: Creatine After Training; Creatine Before Training; Creatine Non-Training

SUMMARY:
Creatine supplementation improves measures of muscle accretion and performance compared to placebo during a resistance training program. However, the optimal creatine supplementation protocol for maximizing these improvements is unknown.

DETAILED DESCRIPTION:
Creatine is a naturally occurring nitrogen containing compound endogenously produced in the body through reactions involving the amino acids arginine, glycine and methionine. Alternatively, creatine can be consumed in the diet (primarily from red meat and seafood) or through commercially manufactured creatine. It has been proposed that the strategic ingestion of creatine supplementation may be an important factor to consider during a resistance training program to increase muscle growth and performance. There is evidence that creatine supplementation only on training days has greater muscle benefits compared to placebo in healthy older adults. However, the effects of creatine on training days (compared to creatine on non-training days or placebo) in healthy young adults is unknown. Further, pre- and post-exercise creatine supplementation appears to produce similar muscle benefits (compared to placebo) in healthy older adults. It remains to be determined whether the timing of creatine ingestion (immediately before vs. immediately following training sessions) influences the physiological adaptations from resistance training compared to placebo in young healthy adults. It is also unknown whether differences exist in supplementing with creatine immediately before, during or immediately following resistance training sessions in young healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (performing structured resistance training > 2x/week for ≥ 4 weeks)
* Males and females (age 18-39)

Exclusion Criteria:

* Pregnant or nursing
* Have consumed creatine monohydrate within 30 days prior to the start of the study
* Pre-existing allergies to the placebo

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Body Composition | baseline, week 16
  Whole-body lean mass (kg) using bioelectrical impedance analysis
Muscle Hypertrophy | baseline, week 16
  Muscle thickness of the biceps, triceps, quadriceps, hamstrings and calf muscle using B-mode ultrasound (cm)
Strength | baseline, week 16
  1-repetition maximum leg press and chest press (kg)
Endurance | baseline, week 16
  Repetitions to fatigue for leg press and chest press (total number)
Power | baseline, week 16
  Medicine ball throw (cm)
Hydration | baseline, week 16
  Total body water (kg) using bioelectrical impedance analysis
Power | baseline, weekn 16
  Vertical jump (watts)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Candow, Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - University of Regina, Regina, Saskatchewan
  - University of Regina, Regina

IPD SHARING:
Plan to Share IPD: No